CLINICAL TRIAL: NCT01288521
Title: Utilizing Pharmacogenetics to Predict Drug Interactions in Kidney Transplant Recipients
Brief Title: Pharmacogenetics to Predict Drug Interactions in Kidney Transplant Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sony Tuteja (Other)
Collaborators: American College of Clinical Pharmacy (Other)
Responsible Party: Sponsor-Investigator, Sony Tuteja, Associate, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 200806718
Record Dates: First submitted 2010-02-09; First posted 2011-02-02 (Estimated); Results first posted 2018-03-09 (Actual); Last update posted 2018-03-09 (Actual); Status verified 2018-02

CONDITIONS: Kidney Transplantation
Keywords: kidney transplantation; tacrolimus; P-glycoprotein; ABCB1; genotyping
MeSH Terms: interventions — Tacrolimus; Ketoconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tacrolimus + Ketoconazole, Then Tacrolimus alone (Experimental): Participants first received tacrolimus in combination with with ketoconazole. After a 1-2 week washout they received tacrolimus alone.
  Interventions: Drug: Tacrolimus + Ketoconazole, Then Tacrolimus alone
- Tacrolimus alone, Then Tacrolimus + Ketoconazole (Experimental): The participants first received tacrolimus alone. After a 1-2 week washout period they received tacrolimus in combination with ketoconazole.
  Interventions: Drug: Tacrolimus alone, Then Tacrolimus + Ketoconazole

INTERVENTIONS:
Drug: Tacrolimus + Ketoconazole, Then Tacrolimus alone — Pharmacokinetic profiling of tacrolimus (AUC0-24h) in subjects receiving tacrolimus + ketoconazole 200 mg every 12 hours x 3 doses.
  Other Names: Tacrolimus; Ketoconazole
  Arms: Tacrolimus + Ketoconazole, Then Tacrolimus alone
Drug: Tacrolimus alone, Then Tacrolimus + Ketoconazole — Pharmacokinetic profiling of subjects on a stable dose of tacrolimus (AUC 0-24h)
  Other Names: Tacrolimus; Ketoconazole
  Arms: Tacrolimus alone, Then Tacrolimus + Ketoconazole

SUMMARY:
Solid organ transplant recipients would greatly benefit from pharmacogenetic evaluation since immunosuppressive drug regimens consist of multiple medications with narrow therapeutic ranges and toxic adverse event profiles. Tacrolimus is a potent immunosuppressive agent utilized for rejection prophylaxis. Intensive pharmacokinetic monitoring must be performed following organ transplantation to ensure therapeutic drug concentrations due to its highly variable pharmacokinetics profile and narrow therapeutic index. Tacrolimus is a substrate for CYP450 3A and for the membrane transporter p-glycoprotein (Pgp). Polymorphisms in the gene encoding for CYP3A5 have been extensively studied and have been found to influence the dosing of tacrolimus. The effect of ABCB1 gene polymorphisms (which encodes for Pgp) upon tacrolimus pharmacokinetics has been more difficult to establish.

This study will determine if haplotypes derived from three frequent polymorphisms in the ABCB1 gene (C1236T, G2677T, C3435T) can predict the degree of drug interaction between tacrolimus (CYP3A5/Pgp substrate) and ketoconazole (CYP3A5/Pgp inhibitor) in patients who are CYP3A5 nonexpressors.

This prospective pharmacokinetic and pharmacogenomic study will enroll 20 stable renal transplant recipients with the CYP3A5 *3/*3 genotype and grouped by ABCB1 haplotype (CGC vs TTT). Pharmacokinetics of tacrolimus will be assessed on 2 occasions with and without ketoconazole coadministration separated by 1 week. The order of study occasions will be randomized in a crossover design.

The results of this study may identify a genomic marker for predicting drug-drug interactions. Knowing this information a priori will aid clinicians in modifying drug dosing and alleviate patients of the burden of significant drug toxicities.

DETAILED DESCRIPTION:
Two mL of blood will be obtained for pharmacogenomic screening for CYP3A5 and ABCB1 genotypes. Patients with the CYP3A5*3/*3 genotype will be consented for the pharmacokinetic portion of the study. Volunteers from this patient cohort will participate in 2 overnight visits to the General Clinical Research Center (GCRC).

Patients will report to the GCRC on the evening before each study visit. They will be required to fast from midnight the night before until 1 hour after tacrolimus administration, which will be in the morning approximately at 8 am.

Pharmacokinetics of tacrolimus will be assessed on 2 occasions with and without ketoconazole coadministration separated by 1 week. The order of study occasions will be randomized in a crossover design. Each patient will take their take their usual oral dose of tacrolimus and have whole blood levels obtained immediately before (C0) and at 0.5, 1, 1.5, 2, 3, 4, 6 hours after the tacrolimus dose. They will then receive tacrolimus by intravenous infusion, a therapeutic dose over four hours. The IV dose will take the place of the patients' usual evening dose of tacrolimus. Additional blood will be drawn for tacrolimus at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 18 hours after the intravenous dose. During the ketoconazole visit, tacrolimus doses will be decreased by one-half to account for the drug interaction and avoid potential tacrolimus-induced toxicities. Ketoconazole 200 mg will be administered orally every 12 hours for a total of 3 doses; the first ketoconazole dose will be given 13 hours before tacrolimus administration.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant recipient
* > 6 months posttransplant
* Serum creatinine < 1.6 mg/dL
* Currently taking a stable dose of tacrolims

Exclusion Criteria:

* On medications known to interact with tacrolimus or ketoconazole
* Multi-organ transplant recipient
* Serum creatinine >1.5 mg/dL

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2008-10; Primary Completion 2011-06 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sony Tuteja, PharmD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Kidney transplant recipients were recruited from the transplant clinic from 10/2008 to 6/2010.
Pre-assignment Details: Assignment to the treatment group was based on CYP3A5 genotype and subjects were eligible only if they had the *3/*3 genotype. 22 subjects were consented to participate. Based on genotype, 3 subjects were ineligible to complete the study. Of the 19 eligible subjects, 11 declined to participate. 8 subjects completed the study.
Groups:
- Tacrolimus + Ketoconazole, Then Tacrolimus Alone; Tacrolimus Alone, Then Tacrolimus + Ketoconazole: Randomized, cross over design
  Tacrolimus + Ketoconazole : Pharmacokinetic profiling of tacrolimus (AUC0-24h) in subjects receiving tacrolimus + keotconazole 200 mg every 12 hours x 3 doses.
  Tacrolimus alone : Pharmacokinetic profiling of subjects on a stable dose of tacrolimus (AUC 0-24h)
Period: Overall Study
Arm/Group | Tacrolimus + Ketoconazole, Then Tacrolimus Alone | Tacrolimus Alone, Then Tacrolimus + Ketoconazole
Started | 3 | 5
Completed | 3 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tacrolimus + Ketoconazole, Then Tacrolimus Alone | Tacrolimus Alone, Then Tacrolimus + Ketoconazole | Total
Number analyzed (Participants) | 3 | 5 | 8
Age, Categorical [Count of Participants; unit: Participants] — Information gathered through self-report and medical records review
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 2 | 5 | 7
    >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (12.5) | 57 (5.5) | 55.6 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 2 | 4 | 6
Region of Enrollment [Number; unit: participants]
  United States | 3 | 5 | 8

OUTCOME MEASURES:

1. Primary Outcome: Tacrolimus Bioavailability (F)
Description: Tac bioavailability alone vs. Tac bioavailability with Keto. To determine F we took the ratio of area under the curve of the oral dose divided by the area under the curve of the IV dose. F was determined by fitting a model that considered the plasma concentration of tac with IV vs. oral dosing.
Time Frame: baseline and 2 weeks
Population: Stable kidney transplant recipients
Measure: Mean (Standard Deviation); unit: ratio of oral to IV
Groups:
- Tacrolimus Alone: cross over design
  Tacrolimus alone : Pharmacokinetic profiling of subjects on a stable dose of tacrolimus (AUC 0-24h)
- Tacrolimus + Ketoconazole: Tacrolimus + Ketoconazole : Pharmacokinetic profiling of tacrolimus (AUC0-24h) in subjects receiving tacrolimus + keotconazole 200 mg every 12 hours x 3 doses.
Arm/Group | Tacrolimus Alone | Tacrolimus + Ketoconazole
Number analyzed (Participants) | 8 | 8
ratio of oral to IV | 0.224 (0.107) | 0.681 (0.308)
Statistical Analysis 1: Comparison: Tacrolimus Alone vs Tacrolimus + Ketoconazole; The bioavailability of Tac alone vs. Tac +keto was compared using a general linear model including sex and creatinine clearance as covariates; Test type: Superiority — The null hypothesis is that the tacrolimus biovailability alone is equal to the tacrolimus bioavailability when given with ketoconazole; p = 0.006, Regression, Linear; The bioavailability with Tac alone vs. Tac +keto was compared using linear model adjusting for sex and creatinine clearance

ADVERSE EVENTS:
Time Frame: Data collected over 6 months of the PK intervention
Groups:
- Tacrolimus Alone: Tacrolimus alone : Pharmacokinetic profiling of subjects on a stable dose of tacrolimus (AUC 0-24h)
Arm/Group | Tacrolimus Alone | Tacrolimus + Ketoconazole
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No